CLINICAL TRIAL: NCT02534545
Title: Remote Ischemic Conditioning for Avoiding Recurrence of Ischemic Stroke in Patients With Symptomatic Intracranial Atherosclerotic Stenosis
Brief Title: Remote Ischemic Conditioning for Avoiding Recurrence of Symptomatic Intracranial Atherosclerotic Stenosis (sICAS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ji Xunming,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming,MD,PhD, VP, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RICA
Record Dates: First submitted 2015-08-23; First posted 2015-08-27 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Intracranial Atherosclerosis
Keywords: Intracranial atherosclerotic stenosis; ischemia; remote ischemic conditioning; stroke
MeSH Terms: conditions — Intracranial Arteriosclerosis; Ischemia; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doctormate® (200mmHg) (Experimental): Patients will be treated with Renqiao Remote Ischemic Conditioning Device (Doctormate®) (200mmHg) once daily for 12 months
  Interventions: Device: Doctormate® (200mmHg)
- Doctormate® (60mmHg) (Sham Comparator): Patients will be treated with the Renqiao Remote Ischemic Conditioning Device (Doctormate®) (60mmHg) once daily for 12 months
  Interventions: Device: Doctormate® (60mmHg)

INTERVENTIONS:
Device: Doctormate® (200mmHg) — Limb ischemia was induced by Renqiao Remote Ischemic Conditioning Device (Doctormate®) inflating tourniquets to 200mmHg.
  Arms: Doctormate® (200mmHg)
Device: Doctormate® (60mmHg) — Limb ischemia was induced by Renqiao Remote Ischemic Conditioning Device (Doctormate®) inflating tourniquets to 60mmHg.
  Arms: Doctormate® (60mmHg)

SUMMARY:
The primary objective of the study will be to determine whether remote limb ischemic conditioning (RLIC) compared with sham RLIC (placebo) treatment reduces the 12-month risk of recurrent IS in patients with a recent TIA or IS caused by stenosis of a major intracranial artery.

After screening period, eligible patients will be randomly allocated into 2 groups. In addition, all participants receive an usual clinical therapy.

DETAILED DESCRIPTION:
In this study, Patients in the RLIC group will be treated with Renqiao Remote Ischemic Conditioning Device (Doctormate®) (200mmHg) once daily for 12 months; patients in the sham RLIC group will be treated with the Renqiao Remote Ischemic Conditioning Device (Doctormate®) (60mmHg) once daily for 12 months. In the study, the RLIC treatment will be comprised of 5 cycles of bilateral upper limb ischemia and reperfusion, which will be induced by 2 cuffs placed around the upper arms respectively and inflated to 200mmHg for 5 minutes followed by 5 minutes of reperfusion by cuff deflation. Sham RLIC treatment will be conducted using the same procedure but with a minimal inflation pressure of 60mmHg, which does not result in upper limb ischemia. In addition, all participants will have received their usual drug therapy according to local medical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female with age from 40 to 80 years old.
2. Patients having an ischemic stroke or a TIA prior to randomization.

   * Patient having an ischemic stroke within 30 days with mRS score≤4 at baseline.
   * Patient having a TIA within 15 days with Oxfordshire Community Stroke Project on the basis of age, blood pressure (BP), clinical features, and duration of TIA symptoms (ABCD2) score≥4 at baseline.
3. The entry event is attributed to symptomatic atherosclerotic stenosis (50-99%) in an intracranial qualifying artery (carotid artery, middle cerebral artery (M1), vertebral artery, or basilar artery) that is documented by magnetic resonance angiography (MRA) or computed tomographic angiography (CTA).
4. Informed consent obtained.

Exclusion Criteria:

1. Thrombolytic therapy within 24 hours prior to enrollment.
2. Progressive neurological signs within 24 hours prior to enrollment.
3. Cerebral venous thrombosis/stenosis.
4. Intracranial arterial stenosis due to arterial dissection, Moya Moya disease; any known vasculitic disease; herpes zoster, varicella zoster or other viral vasculopathy; neurosyphilis; any other intracranial infection; any intracranial stenosis associated with cerebrospinal fluid (CSF) pleocytosis; radiation induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; benign angiopathy of central nervous system; post-partum angiopathy; suspected vasospastic process, suspected recanalized embolus.
5. Any of the following unequivocal cardiac source of embolism: rheumatic mitral and or aortic stenosis, prosthetic heart valves, atrial fibrillation, atrial flutter, sick sinus syndrome, left atrial myxoma, patent foramen ovale, left ventricular mural thrombus or valvular vegetation, congestive heart failure, bacterial endocarditis, or any other cardiovascular condition interfering with the participation.
6. Uncontrolled severe hypertension [sitting systolic blood pressure (SBP) >180 mmHg and/or sitting diastolic blood pressure (DBP) >110 mmHg after medication].
7. Patients with abnormal laboratory parameters: aspartate transaminase (AST) and/or alanine transaminase (ALT) >3×upper limit of normal range; creatinine clearance <0.6 ml/s and/or serum creatinine >265 μmol/l (>3.0 mg/dl); platelets <100×109/L.
8. Any intracranial hemorrhage (parenchymal, subarachnoid, subdural, epidural) within 90 days prior to enrollment.
9. Intracranial neoplasm, cerebral aneurysm or arteriovenous malformation.
10. Known retinal hemorrhage or visceral bleeding within 30 days prior to enrollment.
11. Severe hemostatic disorder or severe coagulation dysfunction.
12. Subclavian arterial stenosis≥50% or subclavian steal syndrome.
13. Extracranial stenosis ≥50%.
14. Previous treatment of target lesion with a stent, angioplasty, or other mechanical device, or plan to perform one of these procedures within 12 months after enrollment.
15. Major surgery (including open femoral, aortic, or carotid surgery, cardiac) within previous 30 days or scheduled in the 12 months after enrollment.
16. Contraindication for remote ischemic conditioning: severe soft tissue injury, fracture, or peripheral vascular disease in the upper limbs.
17. Life expectancy<3 years.
18. Pregnant or breast-feeding women.
19. Unwilling to be followed up or poor compliance for treatment.
20. Patients being enrolled or having been enrolled in other clinical trial within 3 months prior to this clinical trial.
21. Patients unsuitable for enrollment in the clinical trial according to investigators decision making.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The time from randomization to the first occurrence of fatal or non-fatal ischemic stroke. | During the first 12 months from randomization.

SECONDARY OUTCOMES:
The time from randomization to the first occurrence of a composite of fatal or non-fatal stroke (ischemic and hemorrhagic), fatal or non-fatal myocardial infarction, and transient ischemic attack (TIA) . | During the first 12 months from randomization.
The time from randomization to the first occurrence of each component of the composite of fatal or non-fatal stroke (ischemic and hemorrhagic), fatal or non-fatal myocardial infarction, and TIA. | During the first 12 months from randomization.
Time to death from all causes from randomization. | During the first 12 months from randomization.

OTHER OUTCOMES:
Scores assessed by National Institutes of Health Stroke Scale(NIHSS) | During the first 12 months from randomization.
Scores assessed by modified Rankin Scale(mRS) | During the first 12 months from randomization.
Scores assessed by Barthel Index(BI). | During the first 12 months from randomization.
Number of participants with abnormal laboratory values | 3 years
Number of participants with adverse events that are related to treatment | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD. PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (50):
- China (50):
  - Wuhu NO.2 People's Hospital, Wuhu, Anhui
  - The Hospital of Shunyi District Beijing, Beijing, Beijing Municipality
  - Beijing Huairou Hospital, Beijing, Beijing Municipality
  - Baoding No.1 Hospital, Baoding, Hebei
  - Cangzhou People Hospital, Cangzhou, Hebei
  - Hebei Province Cangzhou Hospital of Integrated Traditional and Western Medicine, Cangzhou, Hebei
  - Chengde Central Hospital, Chengde, Hebei
  - Handan First Hospital, Handan, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Shijiazhuang The First Hospital, Shijiazhuang, Hebei
  - Shijiazhuang The Third Hospital, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Houspital of Xingtai, Xingtai, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - The First Clinical Hospital affiliated to Harbin Medical University, Harbin, Heilongjiang
  - The Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Luohe Central Hospital, Luohe, Henan
  - Shangqiu First People's Hospital, Shangqiu, Henan
  - Xuchang Central Hospital, Xuchang, Henan
  - Zhumadian Ctentral Hospital, Zhumadian, Henan
  - Technology The Central Hospital of Wuhan, Wuhan, Hubei
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - Changzhou NO.2 People's Hospital, Changzhou, Jiangsu
  - Anshanshi Changda The Hospital, Anshan, Liaoning
  - Chaoyang Central Hospital, Chaoyang, Liaoning
  - Dalian Municipal Central Hospital Affiliated of Dalian Medical University, Dalian, Liaoning
  - Jinzhou Central Hopital, Jinzhou, Liaoning
  - The Third Affiliated Hospital of Liaoning Medical College, Jinzhou, Liaoning
  - The First People's Hospital of Shenyang, Shenyang, Liaoning
  - The General Hospital of Shenyang Military, Shenyang, Liaoning
  - The Peoele's Hospital of Liaoning Province, Shenyang, Liaoning
  - Ankang City Central Hospital, Ankang, Shaanxi
  - Dezhou People's Hospital, Dezhou, Shandong
  - Shengli Oilfield Central Hospital, Dongying, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Rizhao Hospital of Traditional Chinese Medicine, Rizhao, Shandong
  - Affiliated Hospital of Weifang Medical University, Weifang, Shandong
  - Peace Hospital Affiliated to Changzhi Medical College Shanxi Province, Changzhi, Shanxi
  - Fenyang Hospital of Shanxi Medical Unversity, Fenyang, Shanxi
  - First Hospital of Shanxi Medical Unversity, Taiyuan, Shanxi
  - Shanxi College of Traditional Chinese Medicine Hospital, Taiyuan, Shanxi
  - Tianjin 4th Centre Hospital, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Shaoxing Central Hospital, Shaoxing, Zhejiang
  - Zhoushan Putuo Hospital, Zhoushan, Zhejiang
  - Xuanwu Hospital, Capital Medical University, Beijing
  - Beijing Aerospace General Hospital, Beijing
  - Beijing Luhe Hospital, Capital Medical University, Beijing
  - Xiyuan Hospital, China Academy of Chinses Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hou C, Lan J, Lin Y, Song H, Wang Y, Zhao W, Li S, Meng R, Hao J, Ding Y, Chimowitz MI, Fisher M, Hess DC, Liebeskind DS, Hausenloy DJ, Huang J, Li Z, Han X, Yang J, Zhou J, Chen P, Zhu X, Hu P, Pang H, Chen W, Chen H, Li G, Tao D, Yue W, Gao Z, Ji X; RICA investigators. Chronic remote ischaemic conditioning in patients with symptomatic intracranial atherosclerotic stenosis (the RICA trial): a multicentre, randomised, double-blind sham-controlled trial in China. Lancet Neurol. 2022 Dec;21(12):1089-1098. doi: 10.1016/S1474-4422(22)00335-0. Epub 2022 Oct 27. PMID 36354026